CLINICAL TRIAL: NCT01679171
Title: One Year Outcome of Elderly Patients Admitted to an ICU and Mechanically Ventilated
Acronym: SENIOREA
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC-2012-01; B120579-30 (Other: Agence Nationale de la Santé et du Médicament)
Record Dates: First submitted 2012-08-28; First posted 2012-09-05 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Elderly Care
Keywords: Elderly; Intensive care unit; Outcome; Comprehensive geriatric assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Elderly patients are increasingly admitted in the Intensive Care Unit. Short-term outcome (e.g. hospital survival) of an ICU stay is improving in this population but little data have been published on long-term outcome. Beyond survival, outcome assessment in the elderly requires to evaluate several aspects of health: mental status, activity of daily living, pain, depression, frailty… referred by geriatrician as "comprehensive geriatric assessment' (CGA).

The purpose of the SENIOREA study is to evaluate one year outcome of elderly patients mechanically ventilated in the ICU by performing CGA one year after ICU admission. CGA will be performed on the patients' site of living.

This prospective multicentric trial will be conducted over 8 medico-surgical ICUs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 75 or over
2. Admitted in a participating ICU
3. Requiring mechanical ventilation (invasive or non invasive), initiated before ICU admission or during the 48 first hours after admission.

Exclusion Criteria:

1. Non French-speaking person
2. Failure to obtain a consent by persons authorized to do so.
3. Person non-beneficiary of a social security system.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 75 and over admitted in one of the participating ICU and requiring mechanical ventilation will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2015-07-10 (Actual); Study Completion 2015-07-10 (Actual)

PRIMARY OUTCOMES:
One year outcome | 1 year
  Survival and health status will be assessed using comprehensive geriatric assessment (CGA)

SECONDARY OUTCOMES:
Predictors of one-year outcome | one year
  The secondary assessment criteria as predictors of one year outcome will be researched among:
  * CGA on ICU entry (based on family interview)
  * Vitamin D blood concentration on ICU entry
  * SOFA and SAPSII score on ICU entry
  * Duration of organ dysfunction (ventilator support, renal replacement therapy, vasopressor)
  * ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lerolle, Principal Investigator — CHU Angers France
Locations (1):
- Intensive care unit - CHU Angers, Angers, France

REFERENCES:
- [Derived] Demiselle J, Duval G, Hamel JF, Renault A, Bodet-Contentin L, Martin-Lefevre L, Vivier D, Villers D, Lefevre M, Robert R, Markowicz P, Lavoue S, Courte A, Lebas E, Chevalier S, Annweiler C, Lerolle N. Determinants of hospital and one-year mortality among older patients admitted to intensive care units: results from the multicentric SENIOREA cohort. Ann Intensive Care. 2021 Feb 17;11(1):35. doi: 10.1186/s13613-021-00804-w. PMID 33595733